CLINICAL TRIAL: NCT00003454
Title: Phase II Study of Antineoplastons A10 and AS2-1 In Patients With Carcinoma of the Breast
Brief Title: Antineoplaston Therapy in Treating Women With Stage IV Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066486; BC-BR-12 (Other: Burzynski Research Institute)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Stage IV Breast Cancer
Keywords: recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Patients with Stage IV Breast Cancer will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
RATIONALE: Antineoplastons are naturally-occurring substances that may also be made in the laboratory. Antineoplastons may inhibit the growth of cancer cells.

PURPOSE: This phase II trial studies the effectiveness of antineoplaston therapy in treating women who have stage IV breast cancer that has not responded to previous therapy.

DETAILED DESCRIPTION:
OVERVIEW: This is a single arm, open-label study in which patients with Stage IV breast cancer receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues up to12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in patients with Stage IV breast cancer, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in patients with Stage IV breast cancer.
* To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV breast cancer that is unlikely to respond to existing therapy and for which no curative therapy exists

  * Must have failed prior standard therapy
* Measurable disease by MRI or CT scan
* Tumor must be at least 2 cm in the lymph nodes in the head, neck, axillary, inguinal, or femoral areas and at least 0.5 cm in other locations
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal Status:

* Not specified

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* Bilirubin nor greater than 2.5 mg/dL
* SGOT/SGPT no greater than 5 times upper limit of normal
* No hepatic failure

Renal:

* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No chronic heart failure
* No uncontrolled hypertension
* No history of congestive heart failure
* No history of other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No severe lung disease, such as chronic obstructive pulmonary disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No serious medical or psychiatric disorders
* No active infections
* No other serious concurrent disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy, except in patients with disease progression during or after initial therapy
* Recovery from prior immunotherapy
* No concurrent immunomodulating agents

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas), except in patients with disease progression during or after initial therapy
* Recovery from prior chemotherapy
* No concurrent antineoplastic agents

Endocrine therapy:

* At least 12 weeks since prior hormonal therapy, except in patients with disease progression during and after initial therapy
* Concurrent corticosteroids allowed
* Recovery from prior hormonal therapy

Radiotherapy:

* At least 8 weeks since prior radiotherapy and recovered (patients with multiple tumors who have received radiotherapy to some, but not all, tumors may be admitted earlier than 8 weeks)

Surgery:

* Recovered from any prior surgery

Other:

* No prior antineoplaston therapy
* Prior cytodifferentiating agent allowed

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 1996-03-18 (Actual); Primary Completion 2002-12-28 (Actual); Study Completion 2002-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com